CLINICAL TRIAL: NCT03166826
Title: Development of Modified Combined Apgar Scoring System for Evaluation of Infants in the Delivery Room
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Associate Professor, MD,PhD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 4
Record Dates: First submitted 2016-05-11; First posted 2017-05-25 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Neonatal Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Modified Apgar Scoring System — Modified APGAR scoring system

SUMMARY:
Apgar scoring system has been widely used for the evaluation of the infant's postnatal condition. As conventional Apgar scoring system is affected by gestational age and resuscitative efforts, there is a need for development of new scoring systems for the assessment in the delivery room. Herein, Modified Combined Apgar scoring system which includes two new parameters (cord blood pH and targeted oxygen saturation level) has been developed and the utility of this modified system was compared with Conventional and Combined Apgar scoring systems for prediction of hospitalization.

DETAILED DESCRIPTION:
This is a prospective cohort study. Conventional, Combined and Modified Combined Apgar scores at minutes 1 and 5 are all recorded. For Modified scoring system, blood sample is obtained from the umbilical artery and pulse oximetry is used for measurement of oxygen saturation. Prediction of NICU hospitalization is used as a surrogate parameter to compare the scores.

ELIGIBILITY:
Inclusion Criteria:

Term neonates Preterm neonates Parental approval

Exclusion Criteria :

Major congenital/chromosomal abnormalities Lack of informed consent Stillbirth Outborn infants

Max Age: 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and Preterm Neonates delivered in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Modified Combined Apgar scoring | 10 months
  The predictive value of Modified Combined Apgar scoring for hospitalization of infants

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yilmaz Semerci, MD, Study Director — Kanuni Sultan Suleyman Training and Research Hospital; Gokhan Buyukkale, MD, Study Director — Neonatologist
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No